CLINICAL TRIAL: NCT07018661
Title: [18F]F-FAPI PET/CT and LAparoscopy in STagIng Advanced Gastric Cancer - a Multicenter Prospective Study
Brief Title: [18F]F-FAPI PET/CT and Laparoscopy in Staging Advanced Gastric Cancer
Acronym: PLASTIC-3
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Lioe-Fee de Geus-Oei, MD PhD, Prof. dr., Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 134826; 2024-513255-32-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-04; First posted 2025-06-12 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Gastric Adenocarcinoma; STOMACH NEOPLASM; Gastric Cancer; PET-CT
Keywords: FAPI; 18F-FAPI-74; PET/CT; Imaging biomarker; Gastrectomy; Gastric Cancer; Diagnostics
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]-FAPI-74 PET/CT (Experimental): 3.0 MBq [18F]-FAPI-74 will be administered intravenously 60 minutes before PET/CT scanning. Scanning time will be dependent on the type of scanner in the participating center, but will take approximately 20 minutes.
  Interventions: Diagnostic Test: [18F]FAPI-74 PET/CT; Drug: [18F]-FAPI-74

INTERVENTIONS:
Diagnostic Test: [18F]FAPI-74 PET/CT — Patients included in the study will undergo FAPI-PET/CT after initial staging with gastroscopy and a contrast-enhanced CT of thorax and abdomen, but before undergoing a staging laparoscopy. Based on the results of the FAPI-PET/CT, the MDT and/or treating physician will decide on the next step: confirming possible malignant lesions on PET/CT by biopsies (either percutaneous of by staging laparoscopy), or in case of negative PET/CT, diagnostic laparoscopy.
Drug: [18F]-FAPI-74 — [18F]-FAPI-74 will be administered intravenously 60 minutes before PET/CT-scanning to be able to detect (metastases of) gastric cancer

SUMMARY:
The goal of this clinical trial is to learn if a new type of scan, FAPI-PET/CT, can help find metastases of gastric cancer. We want to know how well this scan works for this purpose and whether it is less burdensome for patients compared to the methods we currently use to find metastases.

The main questions it aims to answer are:

* In how many patients can FAPI-PET/CT find metastases, which leads to a change in their treatment plan as decided by their medical team, such as avoiding unnecessary surgeries and changing from treatment meant to cure the disease to treatment focused on comfort (palliative treatment)?
* In how many patients does FAPI-PET/CT change the diagnostic process as decided by their medical team, like more biopsies or imaging, or changing the type (extent) of surgery needed?

Apart from the usual care gastric cancer patients receive, participants will:

* Undergo one additional scan, which will take approximately 2 hours in total (excluding travel time)
* Complete a number of questionnaires, which will take approximately 4 hours in total

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the stomach or the esophagogastric junction (Siewert type III), by gastroscopy;
* Age greater than or equal to 18 years;
* Surgically resectable, advanced tumor (cT3-4b, N0-3, M0), as determined on gastroscopy and a contrast-enhanced CT of thorax and abdomen. Intention to perform a gastrectomy, based on a multidisciplinary team meeting and shared decision making;
* Patients must have given written informed consent;
* Patients who have recently participated in an interventional study with an investigational medicinal product (IMP) may only participate if an interaction with study procedures is deemed unlikely by the study team (e.g. based on mechanism or washout period).

Exclusion Criteria:

* Siewert type I-II esophagogastric junction tumor;
* Unfit or unwilling to undergo study procedures;
* Unfit or unwilling to undergo surgery;
* Pregnancy at time of the [18F]AlF-FAPI-74 PET/CT scan, due to the investigational PET radiation burden;
* Incapacitated subjects without decision-making capacity;
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent;
* Illiterate patients unable to complete the resource use and quality of life questionnaires;
* Inability to undergo PET/CT scans due to factors such as claustrophobia, weight limits, or the inability to lie flat for the duration of the scan (approximately 30 minutes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in treatment intent | For each patient from enrollment through study completion, an average of 1 year.
  Proportion of patients in whom [18F]AlF-FAPI-74 PET/CT leads to detection of M1-disease resulting in change in treatment intent determined by the local multidisciplinary team (MDT) meetings, including:
  * The number of prevented unnecessary surgeries (staging laparoscopies and/or gastrectomies)
  * The number of changes from curative to palliative treatment
Change in diagnostic work-up | Immediately after completion of clinical staging. Clinical staging consists of FAPI-PET/CT, additional diagnostics following FAPI-PET/CT (if necessary to confirm suspect lesions on FAPI-PET/CT) and/or diagnostic laparoscopy
  Proportion of patients in whom [18F]AlF-FAPI-74 PET/CT leads to changes in diagnostic work-up determined by the local MDT meetings, including:
  * The number of additional biopsies or longitudinal imaging
  * The number of changes in extent of surgery

SECONDARY OUTCOMES:
Diagnostic performance | Immediately after completion of clinical staging. Clinical staging consists of FAPI-PET/CT, additional diagnostics following FAPI-PET/CT (if necessary to confirm suspect lesions on FAPI-PET/CT) and/or diagnostic laparoscopy
  Diagnostic performance measured in sensitivity, specificity, diagnostic accuracy, positive predictive value and negative predictive value using histopathologic tumor tissue collected during biopsy, staging laparoscopy and follow-up imaging as reference test
Incidental findings | Immediately after completion of clinical staging. Clinical staging consists of FAPI-PET/CT, additional diagnostics following FAPI-PET/CT (if necessary to confirm suspect lesions on FAPI-PET/CT) and/or diagnostic laparoscopy
  Proportion of patients with relevant incidental findings (e.g. second primary tumors)
Impact of incidental and/or non-specific findings | At enrollment, after completion of clinical staging but before starting treatment, after completion of clinical staging at 3, 6, 9 and 12 months]
  Patients' extra burden of undergoing additional diagnostics due to incidental and/or non-specific [18F]AlF-FAPI-74 PET/CT findings using EORTC-QLQ-C30. This includes five functional scales, three symptom scales, a global health status/QoL scale and six single items. All of the scales and single-item measures range in score from 0 to 100.
  A high score for a functional scale represents a high/healthy level of functioning.
  A high score for the global health status / QoL represents a high QoL. A high score for a symptom scale/item represents a high level of symptomatology/problems.
Impact of incidental and/or non-specific findings | At enrollment, after completion of clinical staging but before starting treatment, after completion of clinical staging at 3, 6, 9 and 12 months]
  Patients' extra burden of undergoing additional diagnostics due to incidental and/or non-specific [18F]AlF-FAPI-74 PET/CT findings using EQ-5D-5L. This comprises 5 dimensions and each dimension has five response levels, from no problems to unable to/extreme problems. Health states can be summarised using a 5 digit code (one digit for each dimension, no problems is coded as one and extreme problems as 5 and everything in between, e.g. 21111) or represented by a single summary number (index value), through which QALY's can be calculated. The index is derived by applying a formula that attaches values (weights) to each of the levels in each dimension.
Impact of incidental and/or non-specific findings | Immediately after completion of clinical staging. Clinical staging consists of FAPI-PET/CT, additional diagnostics following FAPI-PET/CT (if necessary to confirm suspect lesions on FAPI-PET/CT) and/or diagnostic laparoscopy.
  Patients' extra burden of undergoing additional diagnostics due to incidental and/or non-specific [18F]AlF-FAPI-74 PET/CT findings using a Patient Reported Experience Measure (PREM) questionnaire. This includes questions designed to capture the differences in patient burden between imaging with FAPI-PET/CT and staging laparoscopy. The scale ranges from 1 (strongly agree/not annoying at all) to 5 (strongly disagree/very annoying). A higher score represents a worse outcome.
Diagnostic time delay due to extra investigation | Immediately after completion of clinical staging (after post-diagnostic MDT). Clinical staging consists of FAPI-PET/CT, additional diagnostics following FAPI-PET/CT (if necessary to confirm suspect lesions on FAPI-PET/CT) and/or diagnostic laparoscopy.
  Time between pre-diagnostic and post-diagnostic MDT meetings
Safety data regarding clinical use of [18F]FAPI-74 PET/CT | From start of injection of [18F]FAPI-74 up to 24 hours after administration.
  The occurrence, type, and severity of (serious) adverse events
FAPI-PET based PCI scores | Immediately after staging laparoscopy, which takes place after FAPI-PET/CT.
  Correlation between [18F]AlF-FAPI-74 PET-based Peritoneal Cancer Index (PCI) scores and staging laparoscopy based PCI scores as a reference standard for 'true' intraperitoneal tumor load (this is done only for the LUMC patients).
FAPI uptake and histopathological tumor scores | Immediately after staging laparoscopy
  Correlation between PCI-regional FAPI uptake and PCI-regional histopathological tumor scores (this is done only for LUMC patients).
FAP-expression | Baseline, before study procedure (for D1D2/CRITICS samples) and immediately after gastrectomy or immediately after staging laparoscopy (if no gastrectomy is performed, for PLASTIC-3 patients)
  Expression of CAF content as measured by tumor-stroma ratio (TSR) on tissue samples from D1D2/CRITICS and relation with FAP expression. TSR according to van Pelt and Mesker et al.
TSR, FAP expression and FAPI-PET/CT signals | Immediately after gastrectomy or immediately after staging laparoscopy (if no gastrectomy is performed)
  Analysis of TSR and FAP expression and correlation to [18F]AlF-FAPI-74 PET/CT signal
FAP expressing CAF subsets | Immediately after gastrectomy or immediately after staging laparoscopy (if no gastrectomy is performed)
  Analysis of all FAP expressing CAF subsets in obtained patient samples using imaging mass cytometry
Patient burden | Immediately after completion of clinical staging (after post-diagnostic MDT). Clinical staging consists of FAPI-PET/CT, additional diagnostics following FAPI-PET/CT (if necessary to confirm suspect lesions on FAPI-PET/CT) and/or diagnostic laparoscopy.
  Patient burden using a developed patient reported experience measure (PREM) questionnaire
Health-related quality of life | At enrollment, after completion of clinical staging but before starting treatment, after completion of clinical staging at 3, 6, 9 and 12 months
  Quality of life as measured using the EORTC-QLQ-C30 questionnaire and compared to PLASTIC. The EORTC-QLQ-C30 includes five functional scales, three symptom scales, a global health status/QoL scale and six single items. All of the scales and single-item measures range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status / QoL represents a high QoL. A high score for a symptom scale/item represents a high level of symptomatology/problems.
Health-related quality of life | At enrollment, after completion of clinical staging but before starting treatment, after completion of clinical staging at 3, 6, 9 and 12 months
  Quality of life as measured using the EQ-5D5L questionnaire and compared to PLASTIC. This comprises 5 dimensions and each dimension has five response levels, from no problems to unable to/extreme problems. Health states can be summarised using a 5 digit code (one digit for each dimension, no problems is coded as one and extreme problems as 5 and everything in between, e.g. 21111) or represented by a single summary number (index value), through which QALY's can be calculated. The index is derived by applying a formula that attaches values (weights) to each of the levels in each dimension.
Costs of [18F]FAPI-74 PET/CT | At 3 and 12 months after completion of clinical staging
  Costs of [18F]AlF- FAPI-74 PET/CT compared with staging laparoscopy compared to PLASTIC for patients who received SL only, using the SL bottom-costing approach numbers from the PLASTIC-cost analysis study and resource use questionnaires

CONTACTS AND LOCATIONS:
Locations (10):
- Netherlands (10):
  - ZGT, Almelo
  - Amsterdam UMC, Amsterdam
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam
  - Rijnstate, Arnhem
  - Catharina Ziekenhuis, Eindhoven
  - Zuyderland, Geleen
  - UMC Groningen, Groningen
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification, and only of participants who have given informed consent to share their data for other research purposes will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Investigators with an approved proposal by a review committee may be granted access to research data upon reasonable request, provided necessary privacy provisions are in place. Only data from participants who have given informed consent for its use in other research is included.

REFERENCES:
- [Derived] Triemstra L, Spruijt SWJM, Vriens D, Vegt E, Mesker WE, Hawinkels LJAC, Saing S, Slingerland M, Kemp V, Crobach SALP, Goeman JJ, Pool M, Dibbets-Schneider P, Bennink RJ, van Berge Henegouwen MI, van Det MJ, van Etten BJ, Hartgrink HH, van Hillegersberg R, Lam MGEH, Smulders NM, Luyer MDP, Noordzij W, Owers EC, Oyen WJG, van Sandick JW, Schreurs W, de Steur WO, Stoot JHMB, Weijs LE, Wijnhoven BPL, Witteman BPL, Ruurda JP, de Geus-Oei LF; PLASTIC-3 Study Group. [18F]F-FAPI PET/CT and LAparoscopy in STagIng advanced gastric Cancer: a multicenter prospective study (PLASTIC-3 study). BMC Cancer. 2025 Nov 27;26(1):135. doi: 10.1186/s12885-025-15347-7. PMID 41299326